CLINICAL TRIAL: NCT00004339
Title: Study of Tetrathiomolybdate in Patients With Wilson Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1850; UMMC-801; UMICH-FDU000505
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2003-12

CONDITIONS: Wilson Disease
Keywords: Wilson disease; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Hepatolenticular Degeneration; Metabolism, Inborn Errors; Rare Diseases | interventions — tetrathiomolybdate; Trientine

INTERVENTIONS:
Drug: tetrathiomolybdate
Drug: trientine

SUMMARY:
OBJECTIVES:

Evaluate the safety and efficacy of ammonium tetrathiomolybdate alone and compared with trientine therapy as initial treatment in patients with Wilson disease presenting neurologically.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This a double blind, randomized study. Patients are randomized into one of two treatment arms.

Arm I: Patients receive tetrathiomolybdate (TM) 3 times a day with meals and 3 times a day between meals for 8 weeks in the absence of neurologic deterioration or unacceptable toxicity.

Arm II: Patients receive trientine therapy for 8 weeks in the absence of neurologic deterioration and unacceptable toxicity.

Additional therapy (off study): Patients in the TM group may receive maintenance zinc, while those in the trientine group may continue on trientine or switch to zinc.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Wilson disease presenting with neurologic or psychiatric symptoms
* No concurrent seizure activity
* No white matter lesions on brain magnetic resonance imaging

--Prior/Concurrent Therapy--

* No more than 2 weeks of prior therapy
* No penicillamine or trientine for longer than 2 weeks

--Patient Characteristics--

* Hepatic: No severe hepatic failure
* Other: No psychiatric or medical contraindication to protocol therapy
* Not pregnant

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1994-01

CONTACTS AND LOCATIONS:
Overall Officials: George J. Brewer, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Brewer GJ, Dick RD, Johnson V, Wang Y, Yuzbasiyan-Gurkan V, Kluin K, Fink JK, Aisen A. Treatment of Wilson's disease with ammonium tetrathiomolybdate. I. Initial therapy in 17 neurologically affected patients. Arch Neurol. 1994 Jun;51(6):545-54. doi: 10.1001/archneur.1994.00540180023009. PMID 8198464
- [Background] Brewer GJ, Johnson V, Dick RD, Kluin KJ, Fink JK, Brunberg JA. Treatment of Wilson disease with ammonium tetrathiomolybdate. II. Initial therapy in 33 neurologically affected patients and follow-up with zinc therapy. Arch Neurol. 1996 Oct;53(10):1017-25. doi: 10.1001/archneur.1996.00550100103019. PMID 8859064
- [Background] Brewer GJ, Askari F, Lorincz MT, Carlson M, Schilsky M, Kluin KJ, Hedera P, Moretti P, Fink JK, Tankanow R, Dick RB, Sitterly J. Treatment of Wilson disease with ammonium tetrathiomolybdate: IV. Comparison of tetrathiomolybdate and trientine in a double-blind study of treatment of the neurologic presentation of Wilson disease. Arch Neurol. 2006 Apr;63(4):521-7. doi: 10.1001/archneur.63.4.521. PMID 16606763